CLINICAL TRIAL: NCT05295693
Title: Comparison of the Point-of-care Coagulation Device Quantra With the TEG for Congenital Cardiac Surgery - a Pilot Validation Study
Brief Title: Quantra vs TEG for Congenital Cardiac Surgery - a Pilot Validation Study
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: Quantra vs TEG
Record Dates: First submitted 2022-02-28; First posted 2022-03-25 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Coagulopathy
MeSH Terms: conditions — Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 2 x 2.7mL of full blood for coagulation testing with the Quantra System. Blood samples will not be stored or used for other testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Correlation of the Quantra with the TEG — The purpose of this study is to evaluate the efficacy/reliability/validity of the Quantra device in patients with congenital heart disease for cardiac surgery on CPB.
  The study if of investigational interest only. No clinical decisions will be made based on the results obtained by the Quantra device.

SUMMARY:
Congenital heart surgery on cardio-pulmonary bypass (CPB) is associated with impacted coagulation quality and increased bleeding after separation of CPB.

The current testing device used at our institution is the "TEG 5000" (Haemonetics Corporation). The novel coagulation testing device "Quantra System" (Hemosonics) has favorable properties (result within 20 minutes) allowing for a quicker identification of the coagulation problem and hence faster administration of the correct coagulation products, potentially leading to better coagulation quality and possibly reducing the need of additional blood products. The aim of this prospective observational (non-interventional, investigational only) quality improvement study is to investigate if the Quantra is reliable and valid in predicting the coagulation status when compared with our standard-of-care device TEG 5000.

DETAILED DESCRIPTION:
Congenital heart surgery on cardio-pulmonary bypass (CPB) is associated with impacted coagulation quality and increased bleeding after separation of CPB. Therefore, coagulation products and blood products often need to be given/transfused during these cases. The correct choice and dosing of coagulation products is essential to effectively stop bleeding and reduce the need of additional blood transfusion.

The current testing device used at our institution during congenital heart surgery on CPB is the TEG 5000 (Haemonetics Corporation). Prior to separation from CPB (mostly 30-60 minutes) and after the first coagulation products were given (approx. 60 minutes after separation from CPB) a Clauss Fibrinogen and a TEG are drawn. These samples are sent to an off-site lab for processing and time to result ranges from 60-90 minutes. Therefore, results are often not present when needed.

An easy to use point-of-care (POC) test device being readily available in the operation room and allowing for rapid results could result in quicker identification of the coagulation problem and hence allow for faster administration of the correct coagulation products, potentially leading to better coagulation quality and possibly reducing the need of additional blood products.

The Quantra System (Hemosonics) is an easy-to-use, stand-alone device presenting results within 20 minutes. With these properties all above mentioned problems would be addressed. To date the Quantra has not been used and has not been evaluated in patients with congenital heart disease for cardiac surgery on CPB.

The aim of this prospective observational (non-interventional, investigational only) quality improvement study is to investigate if the Quantra is reliable and valid in predicting the coagulation status when compared with our standard-of-care device TEG

All patients who are enrolled in this study will be patients who are scheduled to undergo cardiac surgery and who require a general anesthesia, endotracheal intubation, arterial line placement and coagulation testing as part of standard of care for the surgery.

No patient will have a general anesthesia, endotracheal intubation, arterial line inserted or coagulation testing for research purposes only.

If the family/patient consent to be enrolled in the study the patient will be included in the study. It is standard of care to draw blood samples for coagulation testing (TEG and Clauss Fibrinogen) prior to separation of cardio-pulmonary-bypass (t1) and after the first coagulation products were given (t2), resulting in 2 x 5.4mL of blood.

For testing of efficacy/reliability/validity of the Quantra System we will need to draw additional blood samples (2.7mL) for each time point t1 and t2, resulting in a total of 2 x 2.7mL. These extra 5.4mL of blood drawn during the research portion of this study is additional to what they need for the surgical procedure and is not standard of care.

No clinical decision will be made on the results of the Quantra System. This is an investigational, non-interventional study.

ELIGIBILITY:
Inclusion Criteria:

* All cases with hypothermia (<=30C)

Exclusion Criteria:

* Neonatal/Infant Bloodless surgery
* Bodyweight under 3kg

Max Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients with congenital heart disease scheduled for cardiac surgery on cardio-pulmonary bypass at our institution Age range is 0 to 8 years. There are no enrollment restrictions related to gender or ethnic background.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-10-13 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
Correlation Quantra vs TEG_Fibrinogen_Function1 | 30 minutes during anesthesia, prior to separation from CPB
  Correlation/Linear regression/normal_vs_abnormal of Quantra (FCS) with TEG (K time & alpha angle)
Correlation Quantra vs TEG_Fibrinogen_Function1 | 30 minutes during anesthesia, after coagulation products were given
  Correlation/Linear regression/normal_vs_abnormal of Quantra (FCS) with TEG (K time & alpha angle)
Correlation Quantra vs TEG_Fibrinogen_Function2 | 30 minutes during anesthesia, prior to separation from CPB
  Correlation/Linear regression/normal_vs_abnormal of Quantra (FCS) with Clauss Fibrinogen.
Correlation Quantra vs TEG_Fibrinogen_Function2 | 30 minutes during anesthesia, after coagulation products were given
  Correlation/Linear regression/normal_vs_abnormal of Quantra (FCS) with Clauss Fibrinogen.
Correlation Quantra vs TEG_Platelet_Function | 30 minutes during anesthesia, prior to separation from CPB
  Correlation/Linear regression/normal_vs_abnormal of Quantra (CS/PCS) with TEG (MA)
Correlation Quantra vs TEG_Platelet_Function | 30 minutes during anesthesia, after coagulation products were given
  Correlation/Linear regression/normal_vs_abnormal of Quantra (CS/PCS) with TEG (MA)
Correlation Quantra vs TEG_clot initiation | 30 minutes during anesthesia, prior to separation from CPB
  Correlation/Linear regression/normal_vs_abnormal of Quantra (CT/CTH) with TEG (R time)
Correlation Quantra vs TEG_clot initiation | 30 minutes during anesthesia, after coagulation products were given
  Correlation/Linear regression/normal_vs_abnormal of Quantra (CT/CTH) with TEG (R time)
Correlation Quantra vs TEG_clot strength/firmness | 30 minutes during anesthesia, prior to separation from CPB
  Correlation/Linear regression/normal_vs_abnormal of Quantra (CS) with TEG (G value)
Correlation Quantra vs TEG_clot strength/firmness | 30 minutes during anesthesia, after coagulation products were given
  Correlation/Linear regression/normal_vs_abnormal of Quantra (CS) with TEG (G value)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander R Schmidt, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ochocinski D, Navaratnam M, Babb A, De Souza E, Kamra K, Sleasman JR, Margetson TD, Bhamidipati JK, Ramamoorthy C, Schmidt AR. Comparison of the Point-Of-Care Coagulation Device Quantra With the TEG-5000 for Congenital Cardiac Surgery-A Pilot Study. Paediatr Anaesth. 2025 Jun;35(6):469-480. doi: 10.1111/pan.15097. Epub 2025 Mar 17. PMID 40095320